CLINICAL TRIAL: NCT00021983
Title: Phase I Study of BL22, a Recombinant Immunotoxin for Treatment of CD22+ Leukemias and Lymphomas
Brief Title: Immunotoxin Therapy in Treating Patients With Hairy Cell Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066835; NCI-99-C-0014; NCI-T98-0063; NCT00001792 (obsolete NCT alias)
Record Dates: First submitted 2001-08-10; First posted 2003-12-12 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2006-01

CONDITIONS: Leukemia
Keywords: refractory hairy cell leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Hairy Cell | interventions — RFB4(dsFv)-PE38 recombinant immunotoxin

INTERVENTIONS:
Biological: BL22 immunotoxin

SUMMARY:
RATIONALE: An immunotoxin can locate cancer cells and kill them without harming normal cells. This may be an effective treatment for hairy cell leukemia.

PURPOSE: Phase I trial to study the effectiveness of BL22 immunotoxin in treating patients who have refractory or recurrent hairy cell leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the toxicity and therapeutic efficacy of recombinant BL22 immunotoxin in patients with refractory or recurrent CD22+ hairy cell leukemia.
* Define the pharmacokinetics of this drug, including the terminal elimination serum half-life area under the curve and volume of distribution, in these patients.
* Evaluate the immunogenicity of this drug in these patients.
* Determine the effect of this drug on various components of the circulating cellular immune system in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive recombinant BL22 immunotoxin IV over 30 minutes on days 1, 3, and 5. Treatment repeats at least every 42 days for up to 4 courses in the absence of disease progression and sufficient neutralizing antibodies.

Cohorts of 3-6 patients receive escalating doses of recombinant BL22 immunotoxin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experiences dose-limiting toxicity.

PROJECTED ACCRUAL: A maximum of 46 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed refractory or recurrent hairy cell leukemia

  * Relapsed after less than 2 years of complete remission after purine analog therapy
  * Must have at least one of the following indications for therapy:

    * Progressive or massive splenomegaly
    * Cytopenia defined by the following:

      * Absolute neutrophil count less than 1,000/mm^3 OR
      * Platelet count less than 100,000/mm^3 OR
      * Hemoglobin less than 12 g/dL
    * More than 20,000 hairy cells/mm^3
    * Symptomatic adenopathy
    * Constitutional symptoms including tumor-related fever or bone pain
* Evidence of CD22 positivity by 1 of the following:

  * More than 15% of malignant cells from a site must react with anti-CD22 by immunohistochemistry
  * More than 30% of malignant cells from a site CD22+ by fluorescent-activated cell sorter
  * More than 400 CD22 sites/cell (average) on malignant cells as assessed by radiolabeled anti-CD22 binding
* No CNS disease requiring treatment
* No patients whose serum neutralizes BL22 immunotoxin in tissue culture, due to either antitoxin or antimouse-IgG antibodies

  * No patients whose serum neutralizes more than 75% of the activity of 1 microgram/mL of BL22 immunotoxin

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 6 months

Hematopoietic:

* See Disease Characteristics
* Pancytopenia due to disease allowed

Hepatic:

* ALT and AST less than 2.5 times upper limit of normal (ULN)
* Bilirubin less than 1.5 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL

Pulmonary:

* FEV1 at least 60% of predicted
* DLCO at least 55% of predicted

Other:

* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior bone marrow transplantation allowed
* At least 3 weeks since prior interferon for the malignancy
* More than 3 months since prior monoclonal antibody therapy (e.g., rituximab)

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior cytotoxic chemotherapy for the malignancy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior whole body electron beam radiotherapy for the malignancy
* Radiotherapy within the past 3 weeks allowed provided less than 10% of total bone marrow was treated and patient has measurable disease outside the radiation port

Surgery:

* Not specified

Other:

* At least 3 weeks since prior retinoids for the malignancy
* At least 3 weeks since any other prior systemic therapy for the malignancy
* No concurrent therapeutic warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-12

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kreitman, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Background] Matsushita K, Margulies I, Onda M, Nagata S, Stetler-Stevenson M, Kreitman RJ. Soluble CD22 as a tumor marker for hairy cell leukemia. Blood. 2008 Sep 15;112(6):2272-7. doi: 10.1182/blood-2008-01-131987. Epub 2008 Jul 2. PMID 18596230
- [Background] Kreitman RJ, Squires DR, Stetler-Stevenson M, Noel P, FitzGerald DJ, Wilson WH, Pastan I. Phase I trial of recombinant immunotoxin RFB4(dsFv)-PE38 (BL22) in patients with B-cell malignancies. J Clin Oncol. 2005 Sep 20;23(27):6719-29. doi: 10.1200/JCO.2005.11.437. Epub 2005 Aug 1. PMID 16061911
- [Result] Kreitman RJ, Wilson WH, Bergeron K, Raggio M, Stetler-Stevenson M, FitzGerald DJ, Pastan I. Efficacy of the anti-CD22 recombinant immunotoxin BL22 in chemotherapy-resistant hairy-cell leukemia. N Engl J Med. 2001 Jul 26;345(4):241-7. doi: 10.1056/NEJM200107263450402. PMID 11474661